CLINICAL TRIAL: NCT02986295
Title: Real World Drug-Eluting Stent Prospective, Open, Multi-site, Registry in Korea: BioMimeTM Stent, Ultimaster® Stent vs. Xience® Stent By SMart Angioplastry Research Team (SMARTDESK-MX)
Brief Title: Registry in Korea: BioMimeTM Stent, Ultimaster® Stent vs. Xience® Stent
Acronym: SMARTDESK-MX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hyeon-Cheol Gwon (Other)
Collaborators: Meril Life Sciences Pvt. Ltd. (Industry); Terumo Corporation (Industry)
Responsible Party: Sponsor-Investigator, Hyeon-Cheol Gwon, Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Other Study IDs: 2016-04-059
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Ischemic Heart Disease
Keywords: BioMime, Ultimaster, Ischemic heart disease, DES
MeSH Terms: conditions — Myocardial Ischemia; Dysequilibrium syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- BioMimeTM Stent: No intervention / Ischemic heart disease with percutaneous coronary intervention with BioMimeTM Stent
  Interventions: Device: BioMimeTM Stent, Ultimaster® Stent
- Ultimaster® Stent: No intervention / Ischemic heart disease with percutaneous coronary intervention with Ultimaster® stent
  Interventions: Device: BioMimeTM Stent, Ultimaster® Stent

INTERVENTIONS:
Device: BioMimeTM Stent, Ultimaster® Stent

SUMMARY:
Comparison of safety and long-term effects of BioMimeTM stent and Ultimaster® stent with Xience® stent

DETAILED DESCRIPTION:
A prospective, open, multicenter, and observational study will register and compare Xience® groups treated in institutions such as the BioMime ™, Ultimaster® group prospectively registered from June 2016.

The Xience® group has already been registered in the previous study (SMARTDESK-BX), so BioMimeTM and Ultimaster® only need to be registered. Follow-up will be conducted until December 2019, and e-CRF will be completed by April 2020.

ELIGIBILITY:
Inclusion Criteria:

1. 19 years old or older
2. Clinical evidence of coronary artery disease including asymptomatic ischemia, stable angina pectoris, acute coronary syndrome (unstable angina, non-ST segment elevation myocardial infarction, ST segment elevation myocardial infarction).
3. Vessel diameter 2.25 ~ 3.5mm, stenosis more than 50% (However, the number of blood vessels, the number of lesions, and the lesion length are not limited)
4. Voluntary written consent to participate in the trial

Exclusion Criteria:

1. Within 24 hours before percutaneous coronary intervention, hemodynamic instability or cardiogenic shock
2. Life expectancy within 2 years

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ischemic heart disease with percutaneous coronary intervention with stenting
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-04-01 (Actual); Primary Completion 2019-01-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of 1-year target lesion failure | 1-year
  The incidence of 1-year target lesion failure (combination of cardiac death, target vessel myocardial infarction, and target vessel revascularization).

SECONDARY OUTCOMES:
Incidence of 30-day and 2-year target lesion failure | 30-day and 2-year
Incidence of 30-day, 1-year, and 2-year deaths | 30-day, 1-year, and 2-year
Incidence of 30-day, 1-year, and 2-year cardiac events | 30-day, 1-year, and 2-year
Incidence of 30-day, 1-year, and 2-year myocardial infarction | 30-day, 1-year, and 2-year
Incidence of 30-day, 1-year, and 2-year target vessel myocardial infarction | 30-day, 1-year, and 2-year
Incidence of 30-day, 1-year, and 2-year revascularization | 30-day, 1-year, and 2-year
Incidence of 30-day, 1-year, and 2-year target revascularization | 30-day, 1-year, and 2-year
Incidence of 30-day, 1-year, and 2-year stroke | 30-day, 1-year, and 2-year
Incidence of acute stent thrombosis at 24 hours, subacute stent thrombosis at 30 days, and stent thrombosis at 1 and 2 years | 24 hours, 30 days, 1 and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon Cheol Gwon, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stone GW, Midei M, Newman W, Sanz M, Hermiller JB, Williams J, Farhat N, Mahaffey KW, Cutlip DE, Fitzgerald PJ, Sood P, Su X, Lansky AJ; SPIRIT III Investigators. Comparison of an everolimus-eluting stent and a paclitaxel-eluting stent in patients with coronary artery disease: a randomized trial. JAMA. 2008 Apr 23;299(16):1903-13. doi: 10.1001/jama.299.16.1903. PMID 18430909
- [Background] Bavry AA, Kumbhani DJ, Helton TJ, Borek PP, Mood GR, Bhatt DL. Late thrombosis of drug-eluting stents: a meta-analysis of randomized clinical trials. Am J Med. 2006 Dec;119(12):1056-61. doi: 10.1016/j.amjmed.2006.01.023. PMID 17145250
- [Background] Stettler C, Wandel S, Allemann S, Kastrati A, Morice MC, Schomig A, Pfisterer ME, Stone GW, Leon MB, de Lezo JS, Goy JJ, Park SJ, Sabate M, Suttorp MJ, Kelbaek H, Spaulding C, Menichelli M, Vermeersch P, Dirksen MT, Cervinka P, Petronio AS, Nordmann AJ, Diem P, Meier B, Zwahlen M, Reichenbach S, Trelle S, Windecker S, Juni P. Outcomes associated with drug-eluting and bare-metal stents: a collaborative network meta-analysis. Lancet. 2007 Sep 15;370(9591):937-48. doi: 10.1016/S0140-6736(07)61444-5. PMID 17869634
- [Background] Vlachojannis GJ, Smits PC, Hofma SH, Togni M, Vazquez N, Valdes M, Voudris V, Puricel S, Slagboom T, Goy JJ, den Heijer P, van der Ent M. Long-term clinical outcomes of biodegradable polymer biolimus-eluting stents versus durable polymer everolimus-eluting stents in patients with coronary artery disease: three-year follow-up of the COMPARE II (Abluminal biodegradable polymer biolimus-eluting stent versus durable polymer everolimus-eluting stent) trial. EuroIntervention. 2015 Jul;11(3):272-9. doi: 10.4244/EIJV11I3A53. PMID 26196753
- [Background] Natsuaki M, Kozuma K, Morimoto T, Kadota K, Muramatsu T, Nakagawa Y, Akasaka T, Igarashi K, Tanabe K, Morino Y, Ishikawa T, Nishikawa H, Awata M, Abe M, Okada H, Takatsu Y, Ogata N, Kimura K, Urasawa K, Tarutani Y, Shiode N, Kimura T. Final 3-Year Outcome of a Randomized Trial Comparing Second-Generation Drug-Eluting Stents Using Either Biodegradable Polymer or Durable Polymer: NOBORI Biolimus-Eluting Versus XIENCE/PROMUS Everolimus-Eluting Stent Trial. Circ Cardiovasc Interv. 2015 Oct;8(10):e002817. doi: 10.1161/CIRCINTERVENTIONS.115.002817. PMID 26446596
- [Background] Kang SH, Park KW, Kang DY, Lim WH, Park KT, Han JK, Kang HJ, Koo BK, Oh BH, Park YB, Kandzari DE, Cohen DJ, Hwang SS, Kim HS. Biodegradable-polymer drug-eluting stents vs. bare metal stents vs. durable-polymer drug-eluting stents: a systematic review and Bayesian approach network meta-analysis. Eur Heart J. 2014 May;35(17):1147-58. doi: 10.1093/eurheartj/eht570. Epub 2014 Jan 23. PMID 24459196